CLINICAL TRIAL: NCT02971202
Title: A Novel Cross-sectional Analysis of Insulin Sensitivity Among Adolescents and Young Adults With Type 1 Diabetes, MODY2, and Normal Controls: the Contribution of Hyperinsulinemia vs. Hyperglycemia to Insulin Resistance
Brief Title: Contribution of Hyperinsulinemia vs. Hyperglycemia to Insulin Resistance in Type 1 Diabetes and Maturity Onset Diabetes of the Young, Type 2 (MODY2)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Justin Gregory, Assistant Professor of Pediatrics, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 161504
Record Dates: First submitted 2016-10-27; First posted 2016-11-22 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Type 1 Diabetes Mellitus; Maturity-Onset Diabetes of the Young, Type 2; MODY2; Insulin Resistance
Keywords: o-glcnacylation; hexosamine
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Maturity-Onset Diabetes of the Young, Type 2; Insulin Resistance | interventions — Glucose Clamp Technique; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hyperinsulinemic, euglycemic clamp: T1DM (Other): Participants will undergo an 8-hour hyperinsulinemic, euglycemic clamp to quantify insulin sensitivity at whole-body and tissue-specific levels. The following hormones will be infused in the study:
  * insulin (12 milliunit (mU)/m^2/min [3x basal] for 150 minutes, then 40 mU/m^2/min [10x basal] for 180 minutes)
  * glucagon (0.65 ng/kg/min [1x basal] for 330 minutes)
  * somatostatin (60 ng/kg/min) These infusions will maintain a basal glucagon level and an increased insulin level in the blood that will be equal between all 3 cohorts.
  A variable infusion of 20% dextrose will be used to maintain plasma glucose within the euglycemic range throughout the hyperinsulinemic portion of the clamp. 6,6-H2 glucose will be infused at a low rate (0.033-0.22 µmol/kg/min) to determine glucose flux during the study.
  Interventions: Drug: Hyperinsulinemic, euglycemic clamp; Drug: 20% dextrose
- Hyperinsulinemic, euglycemic clamp:MODY2 (Other): Participants will undergo an 8-hour hyperinsulinemic, euglycemic clamp to quantify insulin sensitivity at whole-body and tissue-specific levels. The following hormones will be infused in the study:
  * insulin (12 mU/m^2/min [3x basal] for 150 minutes, then 40 mU/m^2/min [10x basal] for 180 minutes)
  * glucagon (0.65 ng/kg/min [1x basal] for 330 minutes)
  * somatostatin (60 ng/kg/min) These infusions will maintain a basal glucagon level and an increased insulin level in the blood that will be equal between all 3 cohorts.
  A variable infusion of 20% dextrose will be used to maintain plasma glucose within the euglycemic range throughout the hyperinsulinemic portion of the clamp. 6,6-H2 glucose will be infused at a low rate (0.033-0.22 µmol/kg/min) to determine glucose flux during the study.
  Interventions: Drug: Hyperinsulinemic, euglycemic clamp; Drug: 20% dextrose
- Hyperinsulinemic euglycemic clamp:Control (Other): Participants will undergo an 8-hour hyperinsulinemic, euglycemic clamp to quantify insulin sensitivity at whole-body and tissue-specific levels. The following hormones will be infused in the study:
  * insulin (12 mU/m^2/min [3x basal] for 150 minutes, then 40 mU/m^2/min [10x basal] for 180 minutes)
  * glucagon (0.65 ng/kg/min [1x basal] for 330 minutes)
  * somatostatin (60 ng/kg/min) These infusions will maintain a basal glucagon level and an increased insulin level in the blood that will be equal between all 3 cohorts.
  A variable infusion of 20% dextrose will be used to maintain plasma glucose within the euglycemic range throughout the hyperinsulinemic portion of the clamp. 6,6-H2 glucose will be infused at a low rate (0.033-0.22 µmol/kg/min) to determine glucose flux during the study.
  Interventions: Drug: Hyperinsulinemic, euglycemic clamp; Drug: 20% dextrose

INTERVENTIONS:
Drug: Hyperinsulinemic, euglycemic clamp — Participants will undergo an 8-hour hyperinsulinemic, euglycemic clamp to quantify insulin sensitivity at whole-body and tissue-specific levels. The following hormones will be infused in the study:
  * insulin (12 mU/m^2/min [3x basal] for 150 minutes, then 40 mU/m^2/min [10x basal] for 180 minutes)
  * glucagon (0.65 ng/kg/min [1x basal] for 330 minutes)
  * somatostatin (60 ng/kg/min) These infusions will maintain a basal glucagon level and an increased insulin level in the blood that will be equal between all 3 cohorts.
  Other Names: glucose clamp; pancreatic clamp
Drug: 20% dextrose — A variable infusion of 20% dextrose will be used to maintain plasma glucose within the euglycemic range throughout the hyperinsulinemic portion of the clamp. 6,6-H2 glucose will be infused at a low rate (0.033-0.22 µmol/kg/min) to determine glucose flux during the study.

SUMMARY:
The purpose of this study is to determine the key factors influencing insulin sensitivity in type 1 diabetes (T1DM) and maturity onset diabetes of the young, type 2 (MODY2).

Our study tests the hypothesis that decreased insulin sensitivity is primarily driven by chronically elevated insulin levels in the blood rather than chronic elevations in blood sugar.

DETAILED DESCRIPTION:
This research will determine whether insulin resistance (IR) in T1DM is predominantly an effect of chronic hyperglycemia, as is commonly accepted, or a consequence of iatrogenic hyperinsulinemia in the peripheral circulation, as alternatively hypothesized. IR is a consistent but under-recognized finding in T1DM. Despite its independent contribution to micro- and macrovascular disease, its underlying cause has not been established nor have strategies to mitigate it been developed. This research will also characterize IR in maturity onset diabetes of the young, type 2 (MODY2), a population for whom IR has been inadequately studied to date.

Insulin therapy in T1DM attempts to achieve euglycemia but does so in an "unphysiologic" way, by delivering insulin into the subcutaneous tissue as compared to physiologic delivery directly into the hepatic portal circulation. Although life-saving, peripheral insulin delivery in T1DM results in a loss of the normal insulin distribution; the physiologic state maintains insulin at 3-fold higher concentrations in the portal circulation compared with the peripheral circulation. IR in T1DM could therefore occur in response to peripheral hyperinsulinemia, a mechanism that would protect against hypoglycemia and ensure adequate glucose delivery to the central nervous system.

MODY2 is a condition that results a mutation in the gene encoding glucokinase (GCK), which in turn causes a defect in β-cell sensitivity to glucose due to reduced glucose phosphorylation. This effectively raises the "set point" for insulin secretion in response to increased glycemia. Because MODY2 patients retain pancreatic insulin secretion, they usually require no insulin therapy and have a normal insulin distribution between the portal and peripheral circulations.

We therefore hypothesize that IR in T1DM 1) is a homeostatic response to increased peripheral insulin concentrations resulting from peripheral insulin delivery and not significantly attributable to hyperglycemia and 2) results primarily from peripheral tissue IR (especially muscle) and not primarily from hepatic IR. Further, we anticipate that patients with MODY2, a population that has hyperglycemia without hyperinsulinemia, will have insulin sensitivity similar to that of otherwise healthy, nondiabetic individuals.

To test this hypothesis, the hyperinsulinemic, euglycemic clamp will be used to assess IR in a cross-sectional study of 3 groups of subjects:

1. non-diabetic control subjects,
2. patients with well controlled T1DM, and
3. patients with MODY2

Key metabolic differences between these 3 groups will enable us to parse out the relative contributions of peripheral hyperinsulinemia vs. hyperglycemia to IR in T1DM and MODY2. Further, the proposed research will provide information on whether novel therapeutic strategies to restore the normal portal to peripheral insulin distribution can normalize insulin sensitivity (e.g. hepatopreferential insulin analogs, intraperitoneal insulin delivery).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for all subjects:

- BMI 19-28 kg/m^2

Additional inclusion criteria for T1DM subjects:

* Age 13-51
* T1DM duration 1-20 years
* HbA1c 5.9-8.0%

Additional inclusion criteria for MODY2 subjects:

* age 13-51
* positive GCK genetic sequencing
* HbA1c 5.9-8.0%

Additional inclusion criteria for control subjects:

* age 18-5.1
* HbA1c < 5.5%

Exclusion Criteria:

Exclusion criteria for all subjects:

* severe hypoglycemia (>= 1 episode in the past 3 months or diagnosis of hypoglycemia unawareness)
* diabetes comorbidities (>= 1 trip to emergency department for poor glucose control in the past 6 months, New York Heart Association Class II-IV cardiac functional status, systolic blood pressure > 140 and diastolic blood pressure > 100 mmHg, fasting triglycerides > 400 mg/dL, liver transaminases > 2 times the upper limit of normal, renal transplantation or serum creatinine > 1.5 mg/dL)
* confounding medications (any systemic glucocorticoid, any antipsychotic, atenolol, metoprolol, propranolol, niacin, any thiazide diuretic, any oral contraceptive pill with > 35 mcg ethinyl estradiol, growth hormone, any immunosuppressant, any anti-hypertensive, any-antilipidemic)
* pregnancy
* Tanner stage < 5

Additional exclusion criteria for T1DM subjects

* any diabetes medication except insulin
* fasting c-peptide > 0.7 ng/mL

Ages: 13 Years to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2016-12; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin M Gregory, MD, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analyzed during the current study are available from the corresponding author upon reasonable request. No applicable resources were generated or analyzed during the current study.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Gregory JM, Smith TJ, Slaughter JC, Mason HR, Hughey CC, Smith MS, Kandasamy B, Greeley SAW, Philipson LH, Naylor RN, Letourneau LR, Abumrad NN, Cherrington AD, Moore DJ. Iatrogenic Hyperinsulinemia, Not Hyperglycemia, Drives Insulin Resistance in Type 1 Diabetes as Revealed by Comparison With GCK-MODY (MODY2). Diabetes. 2019 Aug;68(8):1565-1576. doi: 10.2337/db19-0324. Epub 2019 May 15. PMID 31092478

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hyperinsulinemic, Euglycemic Clamp: T1DM | Hyperinsulinemic, Euglycemic Clamp:MODY2 | Hyperinsulinemic Euglycemic Clamp:Control
Started | 12 | 10 | 11
Started Study | 11 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 2 | 0 | 1
Not completed — Pregnancy | 1 | 0 | 0
Not completed — screen fail after consent | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyperinsulinemic, Euglycemic Clamp: T1DM | Hyperinsulinemic, Euglycemic Clamp:MODY2 | Hyperinsulinemic Euglycemic Clamp:Control | Total
Number analyzed (Participants) | 12 | 10 | 11 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 4 | 0 | 5
  Between 18 and 65 years | 11 | 6 | 11 | 28
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 8 | 24
  Male | 5 | 1 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 10 | 11 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 12 | 10 | 9 | 31
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Whole-body Glucose Utilization (Rd)
Description: The primary outcome is the degree to which Rd (determined using isotopic glucose tracer techniques) during maximal insulin stimulation differs between cohorts.
Time Frame: End of clamp study (the study will last 8 hours)
Measure: Mean (95% Confidence Interval); unit: mg/kg FFM/min
Arm/Group | Hyperinsulinemic, Euglycemic Clamp: T1DM | Hyperinsulinemic, Euglycemic Clamp:MODY2 | Hyperinsulinemic Euglycemic Clamp:Control
Number analyzed (Participants) | 10 | 10 | 10
mg/kg FFM/min | 8.5 [6.1 to 10.9] | 11.0 [9.1 to 13.0] | 12.1 [10.3 to 14.0]

2. Secondary Outcome: Hepatic Insulin Sensitivity
Description: Glucose production (Ra) will be determined using stable isotopic tracer techniques. The extent to which Ra is suppressed at the end of 4 1/2 hours (when glucose Ra by liver has been submaximally suppressed) compared to basal (ΔRa) is directly proportional to hepatic insulin sensitivity.
Time Frame: 4 1/2 hours into clamp study
Measure: Mean (95% Confidence Interval); unit: mg/kg FFM/min
Arm/Group | Hyperinsulinemic, Euglycemic Clamp: T1DM | Hyperinsulinemic, Euglycemic Clamp:MODY2 | Hyperinsulinemic Euglycemic Clamp:Control
Number analyzed (Participants) | 10 | 10 | 10
mg/kg FFM/min | 1.9 [1.5 to 2.2] | 2.1 [1.7 to 2.4] | 1.7 [1.4 to 2.0]

3. Secondary Outcome: Adipose Tissue Insulin Sensitivity
Description: Insulin sensitivity at fat is directly proportional to insulin's ability to suppress lipolysis. Thus, we will determine the extent to which submaximal insulin stimulation (4 1/2 hours into the study) suppresses glycerol and non-esterified free fatty acids (NEFAs) compared to baseline. The extent to which these two metabolites are suppressed is directly proportional to insulin sensitivity in adipose tissue. Here the suppression of NEFA is taken as the secondary outcome parameter.
Time Frame: 4 1/2 hours into clamp study
Measure: Mean (95% Confidence Interval); unit: μmol/L
Arm/Group | Hyperinsulinemic, Euglycemic Clamp: T1DM | Hyperinsulinemic, Euglycemic Clamp:MODY2 | Hyperinsulinemic Euglycemic Clamp:Control
Number analyzed (Participants) | 10 | 10 | 10
μmol/L | 122.4 [-54.36 to 299.1] | 382.3 [244.4 to 520.3] | 392.7 [274.4 to 511.1]

ADVERSE EVENTS:
Time Frame: 1 week
Description: per protocol, hyperglycemia and hypoglycemia are not considered adverse events unless serious
Arm/Group | Hyperinsulinemic, Euglycemic Clamp: T1DM | Hyperinsulinemic, Euglycemic Clamp:MODY2 | Hyperinsulinemic Euglycemic Clamp:Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 4/12 | 3/10 | 3/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyperinsulinemic, Euglycemic Clamp: T1DM (N=12) | Hyperinsulinemic, Euglycemic Clamp:MODY2 (N=10) | Hyperinsulinemic Euglycemic Clamp:Control (N=11)
Vasovagal Response (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1)
nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
IV site pain (General disorders) | 0 (0) | 1 (1) | 2 (2)
Swelling at biopsy site (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2)
Redness at biopsy site (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2)
hypotension (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/02/NCT02971202/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT02971202/ICF_001.pdf